CLINICAL TRIAL: NCT02167997
Title: EffectiveNess and SAfety of Small ANeurysm COiling Trial
Acronym: NANO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: Stryker Neurovascular (Industry)
Responsible Party: Principal Investigator, Avery Evans, MD, Professor, Department of Radiology, University of Virginia
Other Study IDs: 17155
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Aneurysm
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To compare the safety and efficacy of treating small aneurysms with coils specially designed for small aneurysms to historically reported rates of safety and efficacy for the treatment of larger aneurysms.

DETAILED DESCRIPTION:
This is a prospective cohort study whereby patients who undergo endovascular treatment with coils for intracranial aneurysms will be studied for initial procedural and 12-18 month post-treatment outcome. The procedural failure rate (defined above) of treating small aneurysms with specially designed coils will be compared to pre-specified historical occurrences. This evaluation will occur within the framework of "non-inferiority" (i.e. comparable success to coiling of large aneurysms).

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with a ruptured or un-ruptured cerebral aneurysm appropriate for endovascular treatment as determined by the neurovascular team (neurosurgeon/neurointerventionalist)
* Patients between (and including) 18 and 90 years of age.
* Patient HUNT AND HESS Grade 0-3.
* Where required, patient has given fully informed consent to endovascular coiling procedure. If patient cannot consent for themselves, appropriate written consent has been sought from their surrogate, or from appropriate power of attorney.
* Aneurysm < 4mm in maximum diameter.
* Patient is willing and able to return for clinical evaluation and follow-up imaging evaluation (angiography or MRA) at both 6-months and 12-18 months after endovascular treatment.
* The aneurysm has not previously been treated (by coiling or clipping).
* A three-dimensional angiogram has been performed.
* Placement of at least one "Nano" coil, at, or at least close to the neck of the aneurysm.

Exclusion Criteria:

* Patient has more than one aneurysm requiring treatment in the current treatment session. If a patient has multiple aneurysms, but only one will be treated at the time of enrollment, they are eligible for the trial. (Additional aneurysms may be treated at a later date, and may be treated with any coil type that the operator chooses).
* Patient has an H&H score of 4 or 5 after subarachnoid hemorrhage (SAH).
* Medical or surgical co-morbidity such that the patient's life expectancy is less than 1 year.
* Less than 80% by length of Stryker endovascular coils are implanted.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cerebral aneurysms less than 4mm
Sampling Method: Non-Probability Sample
Enrollment: 252 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Procedural failure | 18 Months
  Defined as the composite of technical failure (inability to coil the aneurysm), and complication leading to permanent neurologic injury or death. The second primary outcome relates to the long term effectiveness of the procedure, and is defined as freedom from angiographic recurrence within a period of 12-18 months after the index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Avery J Evans, MD, Principal Investigator — University of Virginia
Locations (19):
- United States (17):
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Radiology Imaging Associates, Englewood, Colorado
  - University of Florida, Gainesville, Florida
  - Lyerly Neurosurgery, Affiliate of Baptist Health, Jacksonville, Florida
  - Norton Neuroscience Institute, Louisville, Kentucky
  - Maine Medical Center, Scarborough, Maine
  - University of Massachusettes, Worcester, Massachusetts
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Riverside Research and Discovery- Riverside Health System, Newport News, Virginia
  - Sentara Neuroscience Institute, Virginia Beach, Virginia
  - Swedish Neurosciences Research, Seattle, Washington
  - Aurora Research Institute, Milwaukee, Wisconsin
- Canada (2):
  - CHUM - Hôpital Notre-Dame Hospital, Montreal, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan